CLINICAL TRIAL: NCT01375478
Title: Multicenter REtrospective Study to Evaluate coMpliance to Therapy and Drug survIval of Tocilizumab (TCZ) in patientS With Moderate to Severe actIve rheumatOid Arthritis in routiNe Daily Clinical Practice (REMISSION Study)
Brief Title: An Observational Study of RoActemra/Actemra in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25580
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This open-label, retrospective, observational study will evaluate the compliance to RoActemra/Actemra (tocilizumab) therapy in patients with moderate to severe rheumatoid arthritis. Six months data will be collected from patients records.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, over 18 years of age
* Moderate to severe rheumatoid arthritis
* RoActemra/Actemra treatment must have been initiated 6 months prior to signing the informed consent form

Exclusion Criteria:

* Patients with rheumatic autoimmune disease other than rheumatoid arthritis
* Patients who are not willing to sign the informed consent form
* Patients who participate in interventional trials during the period of this observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who remained under continued RoActemra/Actemra treatment | 6 months

SECONDARY OUTCOMES:
Reasons for withdrawal | 6 months
Frequency of withdrawal | 6 months
Frequency of dose modification | 6 months
Reasons for dose modification | 6 months
Safety: Incidence of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Greece (6):
  - Athens
  - Crete
  - Pátrai
  - Rhodes
  - Thessaloniki
  - Voula